CLINICAL TRIAL: NCT03815006
Title: An Open-label, Multi-centre, Randomised, Parallel Design Study to Assess the Efficacy of Flash Glucose Monitoring in Adults With Sub-optimally Controlled Type 1 Diabetes.
Brief Title: Flash-glucose Monitoring in Sub-optimally Controlled Type 1 Diabetes (FLASH-UK)
Acronym: FLASH-UK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Portsmouth Hospitals NHS Trust (Other Government); University Hospital Birmingham NHS Foundation Trust (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); University of Manchester (Other); Diabetes UK (Other); Clinical Trials Unit, Manchester (Other); BHR Limited (Industry); East Suffolk and North Essex NHS Foundation Trust (Other); The Adam Practice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B00373
Record Dates: First submitted 2019-01-11; First posted 2019-01-24 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Free Style Libre 2 device (Experimental): At the start, a blood sample will be taken for the measurement of HbA1c. Training and education on the use of FSL2 will be provided by the research team. Participants will be advised to use flash glucose monitoring continuously for the next 24 weeks.
  Interventions: Device: Free Style Libre 2
- Self-monitoring of blood glucose (No Intervention): At the start, a blood sample will be taken for the measurement of HbA1c. Masked FSL will be applied for two weeks, during the last two weeks of control period. Education will focus on using fingerstick measurement for treatment optimisation.

INTERVENTIONS:
Device: Free Style Libre 2 — FreeStyle Libre 2 (FSL2) is a novel glucose monitoring device (Flash glucose monitoring) in the form of a disc worn on the arm for 14 days and a hand-held reader which is designed to largely replace the recommended 4-10 painful finger-stick blood glucose tests required each day for the self-management of type 1 diabetes (T1D).
  Arms: Free Style Libre 2 device

SUMMARY:
FreeStyle Libre (FSL2) is a novel glucose monitoring device (Flash glucose monitoring) in the form of a disc worn on the arm for 14 days, and a hand-held reader which is designed to largely replace the recommended 4-10 painful finger-stick blood glucose tests required each day for the self-management of type 1 diabetes. The purpose of this study is to determine whether flash glucose monitoring with FSL2 device will improve HbA1c over 24 weeks compared to self-monitoring of blood glucose in adults and adolescents (16 or older) with sub-optimally controlled (HbA1c 7.5% to 11%) type 1 diabetes.

This is an open-label, multi-centre, randomised, parallel design study, involving a 2-week run-in period, followed by a 24-week study period during which participants will use either FSL2 or continue usual finger-stick glucose monitoring in random order. A total of up to 156

randomised participants from up to 180 recruited aged 16 years and older with T1D on insulin pump therapy or multiple daily injection therapy were recruited through diabetes clinics in participating centres.

Participants will receive appropriate training to maximise the benefits of FSL2 and finger-stick glucose levels in self-management. The primary outcome is the difference in HbA1c between the two groups at 24 weeks. Secondary outcomes are time spent with glucose levels above and below target, as recorded by FSL2, and other flash glucose-based metrics. Impact on quality of life, diabetes distress, mood, needle burden, disordered eating and treatment satisfaction will also be undertaken. Relative cost-effectiveness of FSL2 device compared with self-monitoring will also be assessed from a UK NHS perspective.

DETAILED DESCRIPTION:
Study Design:

An open-label, multi-centre, randomised, parallel study, in adults and adolescents (16 years and older) with type 1 diabetes and sub-optimal glycaemic control (HbA1c 7.5% to 11%), either on insulin pump treatment or multiple daily injections, contrasting flash glucose monitoring using FreeStyle Libre 2 device with traditional finger-stick glucose monitoring for 24 weeks. Expecting approximately 15% to 20% dropout rate recruitment will aim for 180 participants aiming for 156 randomised and 128 completed participants.

Participant Recruitment:

This is a UK multi-centre and recruitment will take place at the following centres:

1. Diabetes Centres within Manchester University Foundation Trust
2. Royal Derby Hospital, Derby
3. Queen Elizabeth Hospital, Birmingham
4. Addenbrookes Hospital, Cambridge
5. Norfolk and Norwich University Hospital, Norwich
6. Queen Alexandra Hospital, Portsmouth
7. Ipswich Hospital
8. The Adam Practice, Dorset

Each centre will aim to recruit between 25 to 30 participants. Additional diabetes centres surrounding above hospitals may act as participant identification centres. Potential participants will be identified by their treating clinicians and invited to contact the research team. They will be sent the study information leaflets and an invitation by post or in-person to join the study by the research team at least one day before the recruitment visit. The study may also be advertised via social media.

After recruitment, consent, subjects will be randomised for 24-weeks home use of flash-glucose monitoring or 24-weeks use finger-stick glucose monitoring.

Study Visits:

The study includes up to 7 visits for participants completing the study. Maximum time in study is 30 weeks. Each study visit can be scheduled with +/- 2 weeks of the planned visit date.

Visit 1: Recruitment Visit and Screening Assessment

Once the participants have agreed to participate in the study, they will be invited for the recruitment visit, and given a participant ID, when the following activities will be performed by the research team:

* written informed consent/assent
* checking inclusion and exclusion criteria
* medical and diabetes history including the presence of diabetes complications and hypoglycaemia burden
* ethnicity, body weight and height measurement; calculation of BMI
* record of current insulin therapy
* urine or blood pregnancy test (females of child-bearing potential)
* record of occupation and educational attainment
* any history of disordered eating or needle phobia
* previous participation in structured education, the status of carb counting, use of bolus calculator

Screening Blood Sampling

Blood samples will be taken to measure HbA1c (measured at the local laboratory if not done within the last two weeks). Renal and Thyroid function will also be evaluated (if not done in last one year). Less than 15 ml of whole blood will be taken from each participant.

Questionnaires at screening

Evaluation of participants' responses in terms of quality of life, diabetes distress, needle burden, disordered eating, depression and diabetes treatment satisfaction using

1. EQ-5DL-5L questionnaire
2. Type 1 Diabetes Distress Scale (DDS),
3. Diabetes fear of injecting and self-testing (D-FISQ) questionnaire,
4. Diabetes Eating Problem Survey (DEPS-R),
5. Diabetes Treatment Satisfaction Questionnaire (DTSQ),
6. Patient Health Questionnaire (PHQ-9) and
7. The Glucose Monitoring Satisfaction Survey (GMSS).
8. Hypoglycaemia burden will be assessed using Clarke questionnaire and Gold score.

Visit 2: Insertion of the blinded glucose monitoring device

Purpose of visit 2 is to insert a blinded glucose monitor (FreeStyle Libre Pro device). The participant will be provided with instructions about using this device for the next two weeks. Visit two may be combined with visit 1.

Visit 3: Adherence assessment, randomisation and the start of study treatment

During Visit 3, participant's adherence/tolerance of using the flash-CGM over preceding 14 days will be assessed. To proceed with the study participant should have worn the blinded glucose monitoring device for at least ten days' during the last 14 days of the run-in period. If the participant fails to demonstrate adherence or develops any significant allergy or intolerance to the glucose sensor, the study will be terminated, and the participant will be removed from the study. Participant randomisation for the treatment intervention will take place during visit 3.

Initiation of study treatment The participant will arrive at the clinical facility or clinic at the agreed time. Body weight measurement will be made. Participants will be provided with necessary training on the use of study devices according to randomisation.

Training session Participants randomised to flash-glucose monitoring arm will receive education and training about insertion and initiation of the sensor as well as how to use flash-glucose monitoring data for treatment optimisation. They will be encouraged to download data at home to identify pattern recognition. This session will be conducted by a professional diabetes educator or a member of the study team. Education will be tailored to meet the needs of the individual. Participants randomised to conventional finger-stick glucose monitoring arm will be encouraged to use finger-stick glucose levels to optimise treatment and will receive education about insulin dose adjustments using finger-stick glucose levels. The study will try to mimic real-life conditions by continuing participants pre-study diabetes treatment unchanged and finger-stick glucose testing frequency as determined by the participant as required. Participants in both arms will also receive training on sick day rules and dealing with hypo and hyperglycaemia. Participants will be provided with a paper diary to collect information about insulin doses and carbohydrate intake in the last three days of each study month.

Visit 4: (+4 weeks since randomisation): Review data and treatment optimisation Purpose of this visit is to review data from Flash-glucose monitoring and finger-stick glucose monitoring to further optimise treatment. Study devices will be downloaded. Information about insulin doses and any adverse events will be collected.

Visit 5: (+12 weeks since randomisation): Review data and treatment optimisation

Purpose of this visit is to review data from Flash-glucose monitoring and finger-stick glucose monitoring to further optimise treatment. Study devices will be downloaded. Information about insulin doses, participant diaries and any adverse events will be collected. A blood sample will be collected for HbA1c.

Visit 6: (+22 weeks since randomisation): Finger-stick glucose monitoring arm only

Participants randomised to finger-stick glucose monitoring arm will have an extra visit ten weeks after visit 5 to insert a blinded glucose sensor for data capture.

Visit 7: (+24 weeks since randomisation): End of randomised study treatment

The participant will be invited to attend the research centre approximately 12 weeks after Visit 5. This would be the end of 24 weeks randomised study period. All study devices will be downloaded. Insulin usage data will be recorded and diaries collected. The participant will have a blood test for the HbA1c. Body weight measurement will be made. The participant will be asked to complete the same questionnaires completed at Visit 1. In addition, participants in the FSL2 arm will be asked to complete a additional questionnaire exploring expectations and experience of using FSL2 during the study. A subset of participants (n=40 aiming for 25 completed questionnaires) in the FSL2 arm and subset of researchers (n=10) will also be asked to complete additional questionnaires to help with the process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* The participant is ≥16 years old
* The participant has type 1 diabetes, as defined by WHO for at least 1 year or is confirmed C-peptide negative if duration of diabetes is < 1 years
* Participant is treated with insulin pump or multiple daily injection for at least 12 weeks and no plans to change treatment modality during next 28 weeks
* The participant is literate in English for safe study conduct
* Screening HbA1c ≥ 7.5% (58.5mmol/mol) and ≤ 11% (97 mmol/mol) based on analysis from local laboratory
* The participant is willing to wear study glucose sensor and scan for glucose levels at regular intervals
* The participant is willing to follow study specific instructions and improve glucose control
* Female participants of child bearing age should be on effective contraception and must have a negative blood or urine pregnancy test at screening.
* The participant adopting a virtual pathway through the trial is able and willing to post study devices, questionnaires and blood collection kits back to the research team or to the laboratory using pre-paid postal services.
* The participant adopting a virtual pathway through the trial has internet connection, appropriate videoconferencing software and supporting devices to undertake video consultations where necessary.

Exclusion Criteria:

Key exclusion criteria:

* Non-type 1 diabetes mellitus including those secondary to chronic disease
* Any other physical disease or people with known severe mental illness (psychotic disorder, bipolar disorder, dementia, substance and alcohol dependence, learning disabilities, depression with active suicidal ideation) which are likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
* Current users of real-time glucose monitoring sensors or flash-glucose monitoring for more than 4 weeks within last 12 weeks
* Current treatment with drugs known to interfere with glucose metabolism, e.g. systemic corticosteroids, SGLT2 inhibitors, GLP-1 agonists, Pramlinatide, non-selective beta-blockers and MAO inhibitors etc.(patients on stable metformin is not an exclusion)
* Known or suspected allergy against insulin
* Severe visual impairment
* Complete loss of hypoglycaemia awareness
* Significant renal impairment eGFR<30 within previous one year or on dialysis or active retinopathy (defined as presence of maculopathy or proliferative changes) as judged by the investigator
* More than one episode of severe hypoglycaemia as defined by American Diabetes Association (30) in preceding 24 weeks

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United Kingdom (8):
  - The Adam Practice, Poole, Dorset
  - College of Medical and Dental Sciences University of Birmingham, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - University Hospitals of Derby and Burton NHS Foundation Trust, Derby
  - Ipswich Hospital, Ipswich
  - Manchester University NHS Foundation Trust, Manchester
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary study manuscript after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 6 months and ending 3 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal not overlapping with any planned secondary publications from the research team.

REFERENCES:
- [Background] Leelarathna L, Wilmot EG. Flash forward: a review of flash glucose monitoring. Diabet Med. 2018 Apr;35(4):472-482. doi: 10.1111/dme.13584. Epub 2018 Feb 27. PMID 29356072
- [Derived] Leelarathna L, Evans ML, Neupane S, Rayman G, Lumley S, Cranston I, Narendran P, Barnard-Kelly K, Sutton CJ, Elliott RA, Taxiarchi VP, Gkountouras G, Burns M, Mubita W, Kanumilli N, Camm M, Thabit H, Wilmot EG; FLASH-UK Trial Study Group. Intermittently Scanned Continuous Glucose Monitoring for Type 1 Diabetes. N Engl J Med. 2022 Oct 20;387(16):1477-1487. doi: 10.1056/NEJMoa2205650. Epub 2022 Oct 5. PMID 36198143
- [Derived] Wilmot EG, Evans M, Barnard-Kelly K, Burns M, Cranston I, Elliott RA, Gkountouras G, Kanumilli N, Krishan A, Kotonya C, Lumley S, Narendran P, Neupane S, Rayman G, Sutton C, Taxiarchi VP, Thabit H, Leelarathna L. Flash glucose monitoring with the FreeStyle Libre 2 compared with self-monitoring of blood glucose in suboptimally controlled type 1 diabetes: the FLASH-UK randomised controlled trial protocol. BMJ Open. 2021 Jul 14;11(7):e050713. doi: 10.1136/bmjopen-2021-050713. PMID 34261691

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Free Style Libre 2 Device | Self-monitoring of Blood Glucose
Started | 78 | 78
Completed | 78 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Free Style Libre 2 Device | Self-monitoring of Blood Glucose | Total
Number analyzed (Participants) | 78 | 78 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (14) | 44 (15) | 44 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 45 | 42 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 77 | 75 | 152
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 78 | 78 | 156
Glycated Haemoglobin levels [Mean (Standard Deviation); unit: mmol/mol] | 71.6 (9.5) | 69.9 (8.5) | 70.8 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Level at 24 Weeks
Description: The primary outcome is difference in HbA1c between the two groups at 24 weeks.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Free Style Libre 2 Device | Self-monitoring of Blood Glucose
Number analyzed (Participants) | 72 | 69
mmol/mol | 62.8 (8.5) | 67.7 (9.8)

2. Secondary Outcome: HbA1c Level at 12 Weeks
Description: This is the difference in HbA1c between the two groups at 12 weeks
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Percentage With HbA1c ≤ 53 mmol/Mol (7.0%) at 12 Weeks
Description: This is the comparison between arms of percentage with HbA1c ≤ 53 mmol/mol (7.0%) at 12 weeks
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Percentage With HbA1c ≤ 53 mmol/Mol (7.0%) at 24 Weeks
Description: This is the comparison between arms of percentage with HbA1c ≤ 53 mmol/mol (7.0%) at 24 weeks
Time Frame: 24 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Sensor Based - Time Spent in the Target Glucose Range Between 3.9 to 10.0 mmol/l
Description: Time spent in the target glucose range between 3.9 to 10.0 mmol/l (70 to 180mg/dl).
Time Frame: 24 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Sensor Based - Time Spent Below Target Glucose (<3.9mmol/l)
Description: Time spent below target glucose (<3.9mmol/l) (<70mg/dl)
Time Frame: 24 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Sensor Based - Time Spent Above Target Glucose (10.0 mmol/l)
Description: Time spent above target glucose (10.0 mmol/l) (180 mg/dl)
Time Frame: 24 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Sensor Based - Average Glucose Levels
Description: Average glucose levels
Time Frame: 24 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Sensor Based - Standard Deviation Glucose Levels
Description: Standard deviation glucose levels
Time Frame: 24 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Sensor Based - Coefficient of Variation Glucose Levels
Description: Coefficient of variation glucose levels
Time Frame: 24 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Sensor Based - Time With Sensor Glucose Levels < 3.5 mmol/l
Description: The time with sensor glucose levels < 3.5 mmol/l (63 mg/dl)
Time Frame: 24 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Sensor Based - Time With Sensor Glucose Levels < 3.5 mmol/l
Description: The time with sensor glucose levels < 3.0 (54mg/dl)
Time Frame: 24 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Sensor Based - Time With Sensor Glucose Levels < 2.8 mmol/l
Description: The time with sensor glucose levels < 2.8 mmol/l (50 mg/dl)
Time Frame: 24 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Sensor Based - Time With Sensor Glucose Levels in the Significant Hyperglycaemia
Description: The time with sensor glucose levels in the significant hyperglycaemia (glucose levels > 16.7 mmol/l) (300mg/dl)
Time Frame: 24 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Sensor Based - AUC of Glucose Below 3.0mmol/l
Description: AUC of glucose below 3.0mmol/l (54mg/dl)
Time Frame: 24 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Total Daily Average Insulin Dose
Description: Comparison between arms of Total daily average insulin dose
Time Frame: 24 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Daily Average Basal Insulin Dose
Description: Comparison between arms of Daily average basal insulin dose
Time Frame: 24 weeks
Reporting Status: Not Posted

18. Secondary Outcome: Daily Average Bolus Dose
Description: Comparison between arms of Daily average bolus dose
Time Frame: 24 weeks
Reporting Status: Not Posted

19. Secondary Outcome: Average Number of Boluses of Rapid Acting Insulin
Description: Average number of boluses of rapid acting insulin per day
Time Frame: 24 weeks
Reporting Status: Not Posted

20. Secondary Outcome: Number of Freestyle Libre Scans Per Day
Description: Number of Freestyle Libre scans per day in the intervention arm only
Time Frame: 24 weeks
Reporting Status: Not Posted

21. Secondary Outcome: Frequency of Severe Hypoglycaemic Episodes
Description: Frequency of severe hypoglycaemic episodes as defined by American Diabetes Association
Time Frame: 24 weeks
Reporting Status: Not Posted

22. Secondary Outcome: Frequency of Significant Ketosis Events
Description: Frequency of significant ketosis events (plasma ketones >3mmol/l)
Time Frame: 24 weeks
Reporting Status: Not Posted

23. Secondary Outcome: Nature and Severity of Other Adverse Events
Description: Nature and severity of other adverse events.
Time Frame: 24 weeks
Reporting Status: Not Posted

24. Secondary Outcome: Type 1 Diabetes Distress Scale Score
Description: Type 1 Diabetes Distress Scale score compared between arms
Time Frame: 24 weeks
Reporting Status: Not Posted

25. Secondary Outcome: EQ-5D-5L Quality of Life Questionnaire Score
Description: EQ-5D-5L Quality of Life questionnaire
Time Frame: 24 weeks
Reporting Status: Not Posted

26. Secondary Outcome: Patient Health Questionnaire Score
Description: Patient Health Questionnaire: score of 5-9 would be minimal symptoms. any score large than 20 would be categorised as severe major depression
Time Frame: 24 weeks
Reporting Status: Not Posted

27. Secondary Outcome: Diabetes Fear of Injecting and Self-Testing Questionnaire Score
Description: Diabetes fear of injecting and self-testing questionnaire: 15 questions, 6 for Fear of Self injecting, 9 for fear of self testing.
Time Frame: 24 weeks
Reporting Status: Not Posted

28. Secondary Outcome: The Revised Diabetes Eating Problem Survey Score
Description: The revised Diabetes Eating Problem Survey
Time Frame: 24 weeks
Reporting Status: Not Posted

29. Secondary Outcome: Average Number of Days of Libre Usage Per Week
Description: Average number of days of usage per week
Time Frame: 24 weeks
Reporting Status: Not Posted

30. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire Score
Description: Diabetes Treatment Satisfaction Questionnaire
Time Frame: 24 weeks
Reporting Status: Not Posted

31. Secondary Outcome: Glucose Monitoring Satisfaction Survey Score
Description: Glucose Monitoring Satisfaction Survey: 15 questions ranging from 1-5.
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Free Style Libre 2 Device | Self-monitoring of Blood Glucose
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/78
Serious Adverse Events (participants affected / at risk) | 2/78 | 2/78
Other Adverse Events (participants affected / at risk) | 1/78 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Free Style Libre 2 Device (N=78) | Self-monitoring of Blood Glucose (N=78)
Hospital admission (Endocrine disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Free Style Libre 2 Device (N=78) | Self-monitoring of Blood Glucose (N=78)
skin reaction due to sensor (Product Issues) | 1 (1) | 0 (0) — skin reaction due to sensor

LIMITATIONS AND CAVEATS:
please see NEJM publication for details https://www.nejm.org/doi/full/10.1056/NEJMoa2205650

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT03815006/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT03815006/SAP_001.pdf